CLINICAL TRIAL: NCT06475755
Title: A Phase II, Prospective, Randomized, Open Label, Multi-center Study of Tislelizumab Combined With Anlotinib and Platinum Doublet Chemotherapy as Neoadjuvant/Adjuvant With Resectable Stage II-IIIB Non-Small Cell Lung Cancer
Brief Title: Neoadjuvant/Adjuvant Tislelizumab Combined With Anlotinib and Platinum Doublet Chemotherapy With Resectable NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.202405-11
Record Dates: First submitted 2024-05-28; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Non-Small Cell Lung Cancer; Anti Angiogenesis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Angiogenesis Inhibitors; tislelizumab; anlotinib; Cisplatin; Carboplatin; Paclitaxel; Albumin-Bound Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab with anlotinib and platinum-based chemotherapy + Adjuvant Tislelizumab (Experimental): Intervention/treatment:
  Tislelizumab 200mg iv，d1，q3w， Anlotinib 10mg，po，qd1-14，q3w， Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1 Carboplatin AUC of 5 on Day 1 of each 3-week cycle Paclitaxel 175mg/m2 on Day 1 of each 3-week cycle(SQ only) Albumin-bound paclitaxel 260mg/m2，on D1 IV infusion Q3W or 130mg/m2 on D1D8 IV infusion Q3W for each cycle(SQ only) Pemetrexed 500 mg/m2 on Day 1 of each 3-week cycle(NSQ only) Adjuvant: 4 weeks(±7 Days) following surgery, participants receive no more than 16 cycles (cycle length: 3 weeks) of Tislelizumab [200 mg, IV; given on cycle day 1].
  Interventions: Drug: Immunochemotherapy combined with antiangiogenic
- Tislelizumab with platinum-based chemotherapy + Adjuvant Tislelizumab (Other): Tislelizumab 200mg iv，d1，q3w， Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1 Carboplatin AUC of 5 on Day 1 of each 3-week cycle Paclitaxel 175mg/m2 on Day 1 of each 3-week cycle(SQ only) Albumin-bound paclitaxel 260mg/m2，on D1 IV infusion Q3W or 130mg/m2 on D1D8 IV infusion Q3W for each cycle(SQ only) Pemetrexed 500 mg/m2 on Day 1 of each 3-week cycle(NSQ only) Adjuvant: 4 weeks(±7 Days) following surgery, participants receive no more than 16 cycles (cycle length: 3 weeks) of Tislelizumab [200 mg, IV; given on cycle day 1].
  Interventions: Drug: Immunochemotherapy

INTERVENTIONS:
Drug: Immunochemotherapy combined with antiangiogenic — neoadjuvant： Tislelizumab 200mg iv，d1，q3w， Anlotinib 10mg，po，qd1-14，q3w， Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1 Carboplatin AUC of 5 on Day 1 of each 3-week cycle Paclitaxel 175mg/m2 on Day 1 of each 3-week cycle(SQ only) Albumin-bound paclitaxel 260mg/m2，on D1 IV infusion Q3W or 130mg/m2 on D1D8 IV infusion Q3W for each cycle(SQ only) Pemetrexed 500 mg/m2 on Day 1 of each 3-week cycle(NSQ only) Adjuvant: 4 weeks(±7 Days) following surgery, participants receive no more than 16 cycles (cycle length: 3 weeks) of Tislelizumab [200 mg, IV; given on cycle day 1].
  Other Names: Tislelizumab; Anlotinib; Cisplatin; Carboplatin; Paclitaxel; Albumin-bound paclitaxel; Pemetrexed
  Arms: Tislelizumab with anlotinib and platinum-based chemotherapy + Adjuvant Tislelizumab
Drug: Immunochemotherapy — neoadjuvant：Tislelizumab 200mg iv，d1，q3w， Cisplatin 75 mg/m^2 by IV infusion Q3W, given on cycle day 1 Carboplatin AUC of 5 on Day 1 of each 3-week cycle Paclitaxel 175mg/m2 on Day 1 of each 3-week cycle(SQ only) Albumin-bound paclitaxel 260mg/m2，on D1 IV infusion Q3W or 130mg/m2 on D1D8 IV infusion Q3W for each cycle(SQ only) Pemetrexed 500 mg/m2 on Day 1 of each 3-week cycle(NSQ only) Adjuvant: 4 weeks(±7 Days) following surgery, participants receive no more than 16 cycles (cycle length: 3 weeks) of Tislelizumab [200 mg, IV; given on cycle day 1].
  Other Names: Tislelizumab; Cisplatin; Carboplatin; Paclitaxel; Albumin-bound paclitaxel; Pemetrexed
  Arms: Tislelizumab with platinum-based chemotherapy + Adjuvant Tislelizumab

SUMMARY:
This is a Phase II, prospective, randomized, open label, controlled, multi-center study, aim to evaluate the activity of Tislelizumab and Anlotinib and chemotherapy compared with Tislelizumab and chemotherapy before surgery, followed by Tislelizumab alone as adjuvant therapy. The primary objective of this study is to evaluate and compare pathological complete response rate(pCR).

ELIGIBILITY:
Inclusion Criteria:

1. aged 18~75 years old
2. histologically confirmed stage IIA to stage IIIB (IIIB term T2/3/4N2) non-small cell lung cancer (staging based on AJCC 9th edition)
3. ECOG PS score of 0-1;
4. patients are asked to provide an archived tumor tissue sample (FFPE tissue block or approximately ≥ 6 freshly cut unstained FFPE sections) and a pathology report of this baseline sample for PD-L1 and other biomarker analysis). Biopsy samples are requested at baseline if there are no available archival samples or samples are unavailable.
5. Adequate organ and marrow function
6. expected survival ≥ 3 months;
7. be evaluated by a thoracic surgeon and confirmed to be eligible for R0 resection for the purpose of radical treatment
8. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 Target Lesion (TL) at baseline

Exclusion Criteria:

1. those with a known history of CNS metastases;
2. patients with EGFR mutations or ALK translocations;
3. those with imaging (CT or MRI) showing tumor invasion of a major blood vessel (e.g., pulmonary artery or superior vena cava) or those with a high likelihood of fatal hemorrhage due to tumor invasion of a major blood vessel during the follow-up study;
4. prior treatment with immune checkpoint inhibitors, including but not limited to anti-CTLA-4, anti-PD-1 and anti-PD-L1 therapeutic antibodies, and OX-40;
5. previous systemic antivascular therapy;
6. current participation in an interventional clinical trial or receipt of another investigational drug or medical intervention within 4 weeks;
7. presence of active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction (or other factors affecting the absorption of oral medications such as inability to swallow, nausea and vomiting, abnormal physiologic function, malabsorption syndrome, etc.) that require clinical intervention
8. the presence of any signs or history of bleeding constitution; the presence of unhealed wounds, ulcers, or fractures in patients who have experienced any bleeding or hemorrhagic event ≥ CTCAE Grade 3 within 4 weeks prior to enrollment;
9. class III-IV congestive heart failure with poorly controlled and clinically significant arrhythmias (including QTcF ≥450ms in men and ≥470ms in women);
10. difficult-to-control hypertension;
11. history of severe allergy to anlotinib or its prophylactic agents;
12. any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient cerebral ischemic attack, that has occurred within 6 months prior to enrollment in therapy
13. patients whose medical history or test results indicate a hereditary predisposition to bleeding or coagulation disorders that may increase the risk of bleeding
14. active autoimmune disease requiring systemic treatment or history of autoimmune disease with potential for relapse
15. patients requiring long-term systemic glucocorticosteroids (patients requiring inhaled or locally injected glucocorticosteroids due to COPD, asthma may be enrolled) or who have received immunosuppressive therapy within 7 days prior to treatment
16. have an active infection requiring treatment or have used systemic anti-infective medications within one week prior to the first dose;
17. a history of interstitial lung disease, non-infectious pneumonia, or poorly controlled disease, including pulmonary fibrosis, acute lung disease
18. a known history of human immunodeficiency virus (HIV) infection, untreated active hepatitis B (defined as HBsAg positivity along with a detectable HBV-DNA copy number greater than 2,000 IU/ml, and active HCV-infected subjects (HCV antibody positivity with HCV-RNA levels above the lower limit of detection);
19. previous allogeneic stem cell transplantation or organ transplantation.
20. have received a live vaccine within 30 days prior to the first dose (Cycle 1, Day 1);
21. pregnant or lactating women;
22. patients with hypersensitivity to the study drug or excipients;
23. history or evidence of disease that may interfere with the results of the trial, prevent the subject from participating in the study in its entirety, abnormal values of therapeutic or laboratory tests, or other conditions that, in the opinion of the investigator, make enrollment inappropriate The investigator believes that there are other potential risks that make participation in the study inappropriate;
24. stage IIIB exclusion of patients with TxN3 non-small cell lung cancer (staging based on AJCC 9th edition);
25. renal insufficiency: routine urinalysis suggestive of urinary protein ≥++ or confirmed 24-hour urinary protein volume ≥1.0 g;
26. patients with central squamous cell carcinoma confirmed by imaging and pathology;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) in Intent-to-Treat (ITT) analysis set | through study completion, an average of 1 year
  pathological complete response (pCR): defined as no residual tumor cells in the surgically resected tumor specimen and all sampled regional lymph nodes after neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Linna Liu, Study Director — Tang-Du Hospital
Locations (1):
- Tangdu Hospital of the Fourth Millitary Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT06475755/Prot_000.pdf